CLINICAL TRIAL: NCT03504683
Title: Effect of Time-Restricted Feeding on 24-hour Glycemic Control, Blood Pressure, and Cardiovascular Disease Risk Factors in Adults With Prediabetes
Brief Title: MEAL TIMING Study: Effect of Time-Restricted Feeding on 24-hour Glycemic Control, Blood Pressure, and Cardiovascular Disease Risk Factors in Adults With Prediabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Courtney M Peterson, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300001180; R01DK118236 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified by fasting insulin. Within the lowest insulin strata, randomization will be further stratified by biological sex.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early TRE (Experimental)
  Interventions: Behavioral: Early TRE
- Mid-day TRE (Experimental)
  Interventions: Behavioral: Mid-day TRE
- Control Schedule (Placebo Comparator)
  Interventions: Behavioral: Control Schedule

INTERVENTIONS:
Behavioral: Early TRE — Eat between 8 am - 3 pm (or 7 am - 2 pm, if an early riser)
  Other Names: eTRE
  Arms: Early TRE
Behavioral: Mid-day TRE — Eat between 1 pm - 8 pm (or 12 pm - 7 pm, if an early riser)
  Other Names: mTRE
  Arms: Mid-day TRE
Behavioral: Control Schedule — Eat between 8 am - 8 pm (or 7 am - 7 pm, if an early riser)
  Arms: Control Schedule

SUMMARY:
One in three American adults have prediabetes, and up to 70% of adults with prediabetes eventually develop type 2 diabetes. With the high cost of treating diabetes, cost-effective approaches are needed to reduce the incidence of diabetes. One new strategy may be to change when people eat. Studies in rodents suggest that a form of intermittent fasting that limits eating to a short time period each day and involves fasting for the rest of the day (time-restricted eating; TRE) improves blood sugar control and cardiovascular health. Preliminary studies suggest that TRE also improves blood sugar, weight loss, and cardiovascular health in humans. This study will be the first full-scale, controlled feeding trial to determine whether TRE can improve 24-hour blood sugar control, 24-hour blood pressure, and cardiovascular disease risk factors even when food intake is matched to the control group. This clinical trial will also determine whether the benefits of TRE depend on the time of day that people eat. Participants will be assigned to one of three groups: (1) 'Early TRE' (eat between ~8 am-3 pm), (2) 'Mid-day TRE' (eat between ~1 pm - 8 pm), or (3) Control Schedule (~8 am - 8 pm) for 8 weeks. All food will be provided and matched between groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-70 years old
* Prediabetic as determined by HbA1c between 5.7-6.4% or fasting glucose between 100-125 mg/dl with HbA1c >= 5.1%
* Fasting insulin less than 100.0 mU/l and, if HbA1c <5.7%, must also have fasting insulin >= 8.0 mU/l
* BMI between 30-60 kg/m^2
* Wake up at a regular time between 5-8 am

Exclusion Criteria:

* Been diagnosed with diabetes or on diabetes medication or any medication known to affect glucose or 24-hour rhythms in blood pressure
* On weight loss medication
* Change in the dosage of a chronic medication within the past 2 months
* Have a clinically significant laboratory abnormality (e.g., abnormal hemoglobin levels)
* Significant gastrointestinal disease, major gastrointestinal surgery, or gallstones
* Significant cardiovascular, renal, cardiac, liver, lung, adrenal, or nervous system disease that might compromise the participant's safety or data validity
* Evidence of cancer (other than non-melanoma skin cancer) within the last 5 years
* Pregnant or breastfeeding
* Diagnosed psychiatric conditions
* Sleep disorder, circadian disorder, or regularly sleep less than 6 hours per night
* Major change in health or medical history in the past 3 months
* Currently perform overnight shift work
* Regularly eat within a <10.5-hour period each day
* Lost or gained more than 4% of weight in the past 2 months
* Traveled more than 2 time zones away in the 2 months prior to enrolling in this study
* Will travel outside the Central time zone in the 2 weeks prior to testing
* Will travel more than 1 time zone away during this study
* Behavioral factors or other circumstances that may make it difficult for you to follow the study requirements

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hour glucose levels | 8 weeks
  Mean 24-hour glucose levels (mg/dl)
Mean 24-hour insulin levels | 8 weeks
  Mean 24-hour insulin levels (mU/l)
Mean 24-hour C-peptide levels | 8 weeks
  Mean 24-hour C-peptide levels (pmol/l). This is also a proxy for total 24-hour insulin secretion.
Insulin sensitivity | 8 weeks
  Mean value of insulin sensitivity (dl/kg/min/μU/ml) across the three identical meal tolerance tests, as measured by the Oral Minimal Model
Beta-cell responsivity index (a measure of beta-cell function) | 8 weeks
  Mean value of beta-cell responsivity across the three identical meal tolerance tests, as measured by the Oral Minimal Model
Glucose AUCs | 8 weeks
  Glucose area-under-the-curve (mg/dl x hr) during each of three identical meal tolerance tests within a 24-hour period
Insulin AUC | 8 weeks
  Insulin area-under-the-curve (mU/l x hr) during each of three identical meal tolerance tests within a 24-hour period
C-peptide AUC | 8 weeks
  C-peptide area-under-the-curve (pmol/l x hr) during each of three identical meal tolerance tests within a 24-hour period
Peak glucose and mean amplitude of glycemic excursions (MAGE) glucose values | 8 weeks
  mg/dl

SECONDARY OUTCOMES:
Mean 24-hour systolic and diastolic blood pressure | 8 weeks
  mmHg
Daily maximum value, minimum value, and amplitude of systolic and diastolic blood pressure | 8 weeks
  mmHg
Percentage of individuals with non-dipping blood pressure phenotypes | 8 weeks
Heart Rate | 8 weeks
  beats per minute
Lipids | 8 weeks
  Total cholesterol (mg/dl), LDL cholesterol (mg/dl), HDL cholesterol (mg/dl), and triglycerides (mg/dl)
High Sensitivity C-Reactive Protein (hs-CRP) | 8 weeks
  mg/l
Cortisol | 8 weeks
  μg/dl
8-isoprostane | 8 weeks
  pg/ml

OTHER OUTCOMES:
Adherence | 8 weeks
  Percent adherence to assigned meal timing group
Body weight | 8 weeks
  Change in body weight (kg) as measured by scale weight
Appetite across the day | 8 weeks
  Subjective appetite as measured by Visual Analog Scales across the waking day
Appetite | 8 weeks
  Subjective appetite as measured by retrospective Visual Analog Scales (VAS)
Appetite and Cravings | 8 weeks
  Subjective appetite and cravings as measured by Likert scales
Eating Self-Efficacy | 8 weeks
  Eating self-efficacy as measured by the Weight Loss Efficacy Lifestyle Questionnaire (WEL-8)
Sleepiness | 8 weeks
  Sleepiness as measured by the Karolinska Sleepiness Scale (KSS) across the waking day
Current and Preferred Eating Times | 8 weeks
  Current and preferred eating times as measured by a custom designed chrononutrition questionnaire
Mood | 8 weeks
  Mood as measured by the Visual Analog Mood Scales (VAMS)
Positive Affect | 8 weeks
  Positive Affect as measured by the PROMIS Positive Affect Short Form (PASF)
Stress | 8 weeks
  Stress as measured by the Perceived Stress Scale (PSS)
Anxiety | 8 weeks
  Anxiety as measured by the General Anxiety Disorder-7 (GAD-7)
Depression | 8 weeks
  Depression as measured by the Patient Health Questionnaire-9 (PHQ-9)
Sleep Quality | 8 weeks
  Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PQSI) (This study will use the Global PQSI score, which ranges from 0-21, where higher values correspond to worse sleep quality.)
Sleep Timing, Duration, and Chronotype | 8 weeks
  Sleep timing and duration as measured by the Munich Chronotype Questionnaire (MCTQ)
Chronotype | 8 weeks
  Chronotype as assessed by the reduced Morningness-Eveningness Questionnaire (rMEQ)
GPAQ | 8 weeks
  Physical activity as assessed by the General Physical Activity Questionnaire (GPAQ)
Exit Interview | 8 weeks
  Qualitative data on experiences with the eating schedules and barriers, facilitators, and satisfaction factors
Sleep timing outcomes | 8 weeks
  Sleep duration, sleep timing, sleep latency, and wake after sleep onset as measured by actigraphy watch. (These all have units of time)
Sleep efficiency and disruption | 8 weeks
  Sleep efficiency (%) and awakenings (no.), as measured by actigraphy watch. (These all have dimensionless units.)
Other sleep outcomes | 8 weeks
  Sleep Fragmentation Index (awakenings per time), as measured by actigraphy watch

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M. Peterson, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States